CLINICAL TRIAL: NCT00279292
Title: Phase III Randomized Placebo Controlled Trial of EUS Guided Celiac Plexus Neurolysis for Pancreatic Cancer Pain
Brief Title: Randomized Trial of EUS Neurolysis in Pancreas Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R03 DK69947 (completed); R03DK069947 (NIH)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Procedure: Celiac Plexus Neurolysis

SUMMARY:
This is a clinical trial to determine more effective methods of controlling the pain in pancreatic cancer. Although narcotic pain medication are effective, they have many side effects and are underutilized due to social stigma and fear of addiction. Celiac plexus neurolysis is a nerve block procedure that has been shown to be effective in uncontrolled clinical trials. We hypothesized that celiac plexus neurolysis plus pain medication will be more effective and have fewer side effects than pain medication alone. We are evaluating the effectiveness of this standard pain medications with or without celiac plexus neurolysis in a randomized controlled trial. One half of the participants will receive pain medications only and the other half will receive pain medications plus neurolysis, delivered via an endoscopic ultrasound device placed in the stomach.

DETAILED DESCRIPTION:
This is a phase III randomized blinded sham controlled trial of endoscopic ultrasound guided celiac plexus neurolysis. Patients with pancreatic cancer who are unresectable and who have significant pain (> 3 on 0-10 scale) will be enrolled. At the time of a staging endoscopic ultrasound, patients will be randomized to celiac neurolysis or sham (injection of same medication into lumen of stomach). Neurolysis will be performed using standard bupivicaine and ethanol. Patients will be followed for at least 3 months for pain, quality of life and narcotic usage.

ELIGIBILITY:
Inclusion Criteria:

3.1 Unresectable (T4 or M1 or non-regional lymph nodes) or inoperable (due to medical comorbidity) carcinoma of the pancreas as determined by CT or EUS. Patients with extensive portal vein or superior mesenteric vein involvement (T3 by 6th Ed. AJCC staging manual) will be included only if the consulting surgeon feels the patients is unresectable based on the CT scan information.

3.2 Presence of mid-abdominal pain ( 3 on VAS scale) at least 2 days per week, lasting at least 1 hour per day.

3.3 No known coagulopathy as measured by Prothrombin time (INR) 1.5. Pre-EUS INR is not required unless clinically indicated due to known warfarin use or suspected coagulopathy.

3.4 Patient must not require more than 2 l/min oxygen supplementation to maintain saturation >90%.

3.5 > 6 months since previous myocardial infarction or angina. 3.6 ≥ 4 weeks since previous surgery. 3.7 No institution or change in chemotherapy or radiotherapy within 7 days prior (or 14 days post) ESU-CPN. See section 7.0 and 7.1 for details of chemotherapy and radiotherapy allowances.

3.8 Platelets ≥ 50,000. Pre-EUS CBC is not required unless clinically indicated due to known or suspected coagulopathy.

3.9 Life expectancy > 3 months 3.10 Signed and dated informed consent.

Exclusion Criteria:

Unable to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment of ethanol injection versus placebo
injection for pain in pancreatic cancer patients at 1 month and 3 months.

SECONDARY OUTCOMES:
To evaluate mortality and surgical morbidity at 1 month and 3 months
To evaluate magnitude of narcotic use after treatment at 1 month and 3 months
To estimate the period of time pain scores will remain below baseline levels
To estimate the effect of treatment on quality of life at 1 month and 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, MD MPH, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida